CLINICAL TRIAL: NCT05733832
Title: A Randomized Trial of Post-Discharge Transitional Care for Patients With Chronic Liver Disease
Brief Title: A Trial of Post-Discharge Transitional Care for Patients With Chronic Liver Disease
Acronym: TLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Orman, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TLC; R01DK132390 (NIH)
Record Dates: First submitted 2023-01-18; First posted 2023-02-17 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: This study is a stepped-wedge randomized trial of 1,000 patients with advanced liver disease at four high-volume centers over 45 months (250 participants/site; <6 participants/site/month) to evaluate the efficacy of the Transitional Liver Clinic (TLC) compared to control. In the stepped-wedge design, all sites provide usual care (control) during the initial 9-month enrollment interval. At each subsequent 9-month interval, one site is randomized via a computer-generated randomization scheme to crossover to implement the TLC, which will continue through the final interval where all sites will have implemented the TLC. All sites enroll for the entire 45 months and thus contribute patients to both the control and TLC groups.
Masking Description: No masking; all sites will start out as control groups and all will eventually cross over to the TLC model. All sites will know into which group their and all other sites are enrolling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients in the usual care arm will receive standard follow-up care from their usual providers based on recommendations made by inpatient providers at the time of discharge from the hospital.
- Transitional Liver Clinic (TLC) (Active Comparator): Enrolled patients discharged during the experimental TLC intervention implementation period will receive a phone call from TLC staff within 2 business days of discharge followed by an in-person or video telehealth clinic visit with a hepatology APP within 14 days of discharge. TLC staff will provide additional care based on individual patient needs during the 30-day transitional period.
  Interventions: Other: Transitional Liver Clinic (TLC)

INTERVENTIONS:
Other: Transitional Liver Clinic (TLC) — Participants in this intervention receive additional attention from their Hepatology providers in terms of an additional call/telemedicine visit and more specific/additional attention from their Hepatology APP (advanced practice provider) based on individual patient needs
  Arms: Transitional Liver Clinic (TLC)

SUMMARY:
Patients with complications of advanced liver disease often have difficulties after hospital discharge that result in early hospital readmission. Poor outcomes for these patients during this transitional time could be improved through the use of innovative transitional care models. This proposal aims to examine the effect of a transitional care model, The Transitional Liver Clinic (TLC), in reducing hospital re-admissions, improving quality of life, and improving patient experience.

DETAILED DESCRIPTION:
This study is a stepped-wedge randomized trial of 1,000 patients with advanced liver disease at four high-volume centers over 45 months (250 participants/site; <6 participants/site/month) to evaluate the efficacy of the Transitional Liver Clinic (TLC) compared to control.

In the stepped-wedge design, all sites provide usual care (control) during the initial 9-month enrollment interval. At each subsequent 9-month interval, one site is randomized via a computer-generated randomization scheme to crossover to implement the TLC, which will continue through the final interval where all sites will have implemented the TLC.

All sites enroll for the entire 45 months and thus contribute patients to both the control and TLC groups. There are an equal number of TLC and control intervals; thus approximately 500 patients will be in each group. Participant follow-up will occur by telephone at 30 and 90 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥18
2. Diagnosis of advanced liver disease, defined as either (must meet either a or b)

   1. cirrhosis based on (either i or ii):

      * biopsy
      * characteristic clinical, laboratory, and imaging findings
   2. acute alcoholic hepatitis, defined by NIAAA Alcoholic Hepatitis Consortia, as

      * onset of jaundice (serum bilirubin >3.0 mg/dL) in prior 8 weeks
      * consumption of >40 (female) or 60 (male) g alcohol/day for ≥6 months, with <60 days abstinence before jaundice onset,
      * AST>50 IU/L, AST/ALT>1.5, and both values <400 IU/L
      * liver biopsy confirmation in patients with confounding factors
3. Has at least one of the following complications due to advanced liver disease occurring during hospitalization:

   1. ascites requiring diuretics or paracentesis
   2. hepatic encephalopathy requiring lactulose or rifaximin
   3. gastrointestinal bleeding due to portal hypertension
   4. jaundice
4. Has planned discharge alive to home or a facility within 72 hours of informed consent
5. Able and willing to provide informed consent

Exclusion Criteria:

1. discharge under hospice
2. listed for liver transplant with MELD-Na ≥ 35
3. unable or unwilling to participate in post-discharge follow-up either in-person or virtually
4. unable to speak or understand English and/or Spanish
5. low hearing or communicative ability (examiner rated) that would interfere with interventions and outcome assessments
6. lack of access to a telephone
7. incarcerated
8. concurrent enrollment in an interventional research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
30-day hospital readmissions for patients hospitalized with complications of advanced liver disease | 30 days after discharge of initial hospitalization at which the participant was enrolled in the study.
  The primary outcome, 30-day hospital readmission, is publicly reported by CMS, and is the benchmark measure in the Hospital Readmissions Reduction Program. It is therefore the most appropriate primary outcome.
Quality of life for patients hospitalized with complications of advanced liver disease via Promis 29+2 survey | 30 days after discharge of initial hospitalization at which the participant was enrolled in the study.
  This measure includes 4 items in each of 7 health domains (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference) as well as a single item assessing pain intensity. Each domain is scored using a T-score metric in which 50 corresponds to the average for the US population with a standard deviation of 10, and a higher T-score represents more of the concept being measured. For example, higher fatigue scores indicate more fatigue (worse quality of life), while higher physical function scores represent better physical function (better quality of life).
Quality of life for patients hospitalized with complications of advanced liver disease via Promis 29+2 survey | 90 days after discharge of initial hospitalization at which the participant was enrolled in the study
  This measure includes 4 items in each of 7 health domains (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference) as well as a single item assessing pain intensity. Each domain is scored using a T-score metric in which 50 corresponds to the average for the US population with a standard deviation of 10, and a higher T-score represents more of the concept being measured. For example, higher fatigue scores indicate more fatigue (worse quality of life), while higher physical function scores represent better physical function (better quality of life).
Patient satisfaction for patients hospitalized with complications of advanced liver disease via the PSQ 18 questionnaire | 30 days after discharge of initial hospitalization at which the participant was enrolled in the study
  The PSQ-18 consists of 18 items examining 7 dimensions of satisfaction with medical care: general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, and accessibility and convenience. Each item is scored with a 1 to 5 Likert scale and the individual item scores are averaged, with higher scores reflecting higher satisfaction.
Patient satisfaction for patients hospitalized with complications of advanced liver disease via the PSQ 18 questionnaire | 90 days after discharge of initial hospitalization at which the participant was enrolled in the study
  The PSQ-18 consists of 18 items examining 7 dimensions of satisfaction with medical care: general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, and accessibility and convenience. Each item is scored with a 1 to 5 Likert scale and the individual item scores are averaged, with higher scores reflecting higher satisfaction.

SECONDARY OUTCOMES:
Number of ER visits | 30 days after discharge of initial hospitalization at which the participant was enrolled in the study and 90 days after discharge of initial hospitalization at which the participant was enrolled in the study
  Recognizing the limitations on CMS data, the number of ER visits for each participant will be taken from the medical record and will be measured as a secondary outcome to provide a fuller picture of acute care utilization.
90 day mortality | 90 days after discharge of initial hospitalization at which the participant was enrolled in the study.
  Recognizing the limitations on CMS data, 90 day mortality will be measured as a secondary outcome to provide a fuller picture of acute care utilization.
Days alive out of the hospital | 90 days after discharge of initial hospitalization at which the participant was enrolled in the study.
  Recognizing the limitations on CMS data, number of days alive out of the hospital will be measured as a secondary outcome to provide a fuller picture of acute care utilization.
Hospital readmissions | 30 days after discharge of initial hospitalization at which the participant was enrolled in the study and 90 days after discharge of initial hospitalization at which the participant was enrolled in the study
  Participants will self report or data will be obtained from local institutional medical records the number of times, if any, they were admitted to the hospital during their time of participation in this study

CONTACTS AND LOCATIONS:
Overall Officials: Eric Orman, MD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Indiana University Division of Gastroenterolgy and Hepatology, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No